CLINICAL TRIAL: NCT04634942
Title: A Comparison of Two dıfferent Methods to Reduce ıntramuscular ınjectıon paın; Cold Spray and ShotBlocker
Brief Title: A Comparison of Two Different Methods to Reduce Intramusculer Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeliha CENGİZ, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020/30
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: Intramuscular Injection; Pain; Cold Spray; ShotBlocker
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: In the study, the randomization method was used to assign the patients to the groups to prevent manipulations that could be done consciously or unconsciously. A computer-assisted randomization program was used to make assignments to the groups. A random list was created in the computer environment by using random.org, assigning individuals to groups (117). 195 people, who will form the sample of the study, were divided into sets of 39, and sets were created by assigning numbers from 1 to 5 to each set. When the sets were obtained, the numbers from 1 to 5 were written on small papers, and group assignments were made by lot method.
  Group 1 = Control Group 2 = Cold Spray Placebo 3rd Group = Cold Spray 4th Group = ShotBlocker Group 5 = ShotBlocker Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cold Spray Group (Experimental): Cold spray group injection process step; In addition to the IM injection procedure steps, Cryos cold spray was applied to patients in this group after skin cleansing. Cryos cold spray sprayed 3 puffs from a distance of 20 cm to the skin, and the injection process was performed. Within 2 minutes after the injection process was completed, the patient was allowed to mark the intensity of pain caused by the needle while entering the tissue on the VAS.
  Interventions: Device: Cryos REF 0971 Cold Spray
- ShotBlocker Group (Experimental): ShotBlocker group injection process step; In addition to the IM injection procedure steps, after cleansing the skin of the patients in this group, the protruding part of the ShotBlocker was placed in contact with the skin. ShotBlocker was pressed firmly against the skin and the injection was made through the central opening of the ShotBlocker. ShotBlocker was removed from the skin after the injection was completed. Within 2 minutes after the injection process was completed, the patient was allowed to mark the intensity of pain caused by the needle while entering the tissue on the VAS.
  Interventions: Device: ShotBlocker BIONIX Press Firmly USA
- Control Group (No Intervention): Control group injection process step; The individuals in this group were injected by following the routine IM injection procedure steps. Within 2 minutes after the injection process was completed, the patient was allowed to mark the intensity of pain caused by the needle entering the tissue on the VAS.
- Cold Spray Placebo Group (Placebo Comparator): Cold spray placebo group injection procedure step; In addition to the IM injection procedure steps, the patients in this group were treated with tap water in a cold spray bottle after cleansing the skin. After spraying 3 puffs of tap water in a placebo bottle at a distance of 20 cm to the skin, the injection was performed. Within 2 minutes after the injection process was completed, the patient was allowed to mark the intensity of pain caused by the needle entering the tissue on the VAS.
  Interventions: Device: Cryos REF 0971 Cold Spray
- ShotBlocker Placebo Group (Placebo Comparator): ShotBlocker placebo group injection procedure step; In addition to the IM injection procedure steps, in patients in this group, the non-protruding part of the ShotBlocker was placed in contact with the skin after skin cleaning. ShotBlocker was pressed firmly against the skin and the injection was applied through the central opening of the ShotBlocker. ShotBlocker was removed from the skin after the injection was completed.
  Interventions: Device: ShotBlocker BIONIX Press Firmly USA

INTERVENTIONS:
Device: Cryos REF 0971 Cold Spray — Cold Spray Coolant spray is manufactured from liquefied gases with high pressure. It acts by rapidly reducing the temperature in the body area where it is applied. The liquefied gas in the tube spreads on the skin in liquid form and takes the heat of the skin by turning into gas. The temperature of the area where it is applied drops from 30-32 degrees to 10-15 degrees. With the effect of the cold, the excitability of the nerve endings decreases, and thus the pain on the skin is felt by the person. Cold sprays, whose analgesic effect occurs immediately, are applied parallel to the muscle fibers in the area to be applied, from a distance of 15-45 centimeters, by squeezing for approximately 5-15 seconds. Cold sprays are suitable for long-term and multiple uses.
  Arms: Cold Spray Group; Cold Spray Placebo Group
Device: ShotBlocker BIONIX Press Firmly USA — ShotBlocker ShotBlocker is a plastic tool with a small and flat shape, with short and non-sharp protrusions on one side that connect with the skin. It resembles a horseshoe (C shaped) with its structure designed to expose the area to be injected. It is suitable for all age groups. It does not have any side effects. ShotBlocker can be used for both intramuscular and subcutaneous injections. The protruding surface of the ShotBlocker is held by pressing the skin during the injection and the process is performed from the part where the opening is.
  Arms: ShotBlocker Group; ShotBlocker Placebo Group

SUMMARY:
When the literature is reviewed, there are few studies evaluating cold spray or ShotBlocker in reducing pain associated with IM injection. Studies have shown that these applications are mostly used in children during vaccination or intravenous interventions. These methods are less commonly used on adults. Both methods without side effects are important in terms of being cheap, easy to use and reusable. As a result of the researches, these methods can provide a more comfortable injection experience and provide evidence for pain management, especially in adults sensitive to pain.

The aim of the study is to use it to reduce pain associated with IM injection in adults.

To evaluate the effect of cold spray and ShotBlocker applications on pain.

DETAILED DESCRIPTION:
When the literature is reviewed, there are few studies evaluating cold spray or ShotBlocker in reducing pain associated with IM injection. Studies have shown that these applications are mostly used in children during vaccination or intravenous interventions. These methods are less commonly used on adults. Both methods without side effects are important in terms of being cheap, easy to use and reusable. As a result of the researches, these methods can provide a more comfortable injection experience and provide evidence for pain management, especially in adults sensitive to pain.

The aim of the study is to use it to reduce pain associated with IM injection in adults.

To evaluate the effect of cold spray and ShotBlocker applications on pain. In this study, it was used to reduce pain associated with IM injection in adults.

It was aimed to evaluate the effect of ShotBlocker and cold spray application on pain. The research is planned to be completed between February 2020 and December 2020. The universe of the study, which was conducted as a randomized controlled trial model, consisted of all adult patients who received diclofenac sodium treatment in Malatya Turgut Özal Medical Center Emergency Service. 195 patients selected by the simple random sampling method (shotBlocker group = 39, shotBlocker placebo = 39 spray groups = 39, spray group placebo = 39, control group = 39) were included in the study. Participant Introduction Form and Visual Benchmarking Scale (VAS) were used to collect data. According to the characteristics of the data In independent groups, t test, ANOVA test, Mann Whitney U test, correlation were measured.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Communication,
* Having no problems with vision and hearing,
* No pain, scar tissue, incision, lipodystrophy and signs of infection in the application area,
* Body mass index between 18.5 and 30,
* There is no history of allergy.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2010-02-25 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
The effect of cold spray on intramuscular pain | About 2 months
  The Visual Benchmark Scale (VAS) is a two-tailed 10 cm long scale used to measure pain, expressed by minimum no pain (0) and maximum very severe pain (10). Within 2 minutes of completing the injection, the individual was asked to mark his pain on the The Visual Benchmark Scale (VAS).
The effect of ShotBlocker on intramuscular pain | About 2 months
  The Visual Benchmark Scale (VAS) is a two-tailed 10 cm long scale used to measure pain, expressed by minimum no pain (0) and maximum very severe pain (10). Within 2 minutes of completing the injection, the individual was asked to mark his pain on the The Visual Benchmark Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Malatya Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This research is a master thesis study. The research will be expected to be completed.